CLINICAL TRIAL: NCT05278091
Title: Evaluation of the Diagnostic Value of Video-oculography in CANVAS (Cerebellar Ataxia With Neuropathy and Vestibular Areflexia Syndrome) Neuronopathies
Brief Title: Evaluation of the Diagnostic Value of Video-oculography in CANVAS Neuronopathies
Acronym: VOG-Neuropat
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2022/II-02
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cerebellar Ataxia
MeSH Terms: conditions — Cerebellar Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with CANVAS with genetic confirmation: Patients with CANVAS with genetic confirmation (RFC1 gene mutation)
  Interventions: Other: None, pure observationnal study
- others patients: Patients with axonal neuropathy, autoimmune neuronopathy and anti-MAG neuropathy
  Interventions: Other: None, pure observationnal study
- Healthy controls: Patients without CANVAS or other neuropathy
  Interventions: Other: None, pure observationnal study

INTERVENTIONS:
Other: None, pure observationnal study — None, pure observationnal study

SUMMARY:
Cerebellar ataxia syndrome with neuropathy and vestibular areflexia (CANVAS) is a genetic pathology of recent discovery (bi-allelic expansion in intron 1 of the RFC1 gene with AAGG repetition). The clinical picture is protean, associating a neuronopathy, a bilateral vestibulopathy evidenced by an alteration of the oculovestibular reflex (VOR), an atrophy of the cerebellum and a chronic cough.

In the initial stage of the disease the clinical picture is heterogeneous and often incomplete. Ataxia at the beginning of the disease may be the consequence of peripheral nervous system involvement (neuronopathy) and the cerebellar syndrome may manifest itself clinically late.

Eye movement involvement in central nervous system pathologies is common (4). Oculomotor abnormalities are often subclinical and sometimes exclusively identifiable by an instrumental study, video-oculography (VOG) (5).

VOG is a non-invasive examination of eye movements, which is increasingly used in the differential diagnosis of neurodegenerative syndromes (6). This examination allows, among other things, to identify oculomotor anomalies, even discrete and asymptomatic, by studying the combined movements of the eyes and the oculocephalic movements.

The study of oculomotricity by VOG can therefore potentially contribute to the early differential diagnosis of ataxiating neuropathies, including CANVAS, by revealing infra-clinical oculomotor abnormalities correlated with a cerebellar expectation (knowing the role of the dorsal vermis in the precision of saccades and pursuits).

ELIGIBILITY:
Inclusion Criteria:

Patients followed at the University Hospital of Nîmes between 2018-2021

* Age > 18 years
* Patients with CANVAS with genetic confirmation (RFC1 gene mutation)
* Patients with axonal neuropathy, autoimmune neuronopathy and anti-MAG neuropathy
* Healthy controls

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients followed at the CHU of Nîmes between 2018-2021, with a diagnosis of CANVAS with several control groups constituted by patients with a neuropathy of different etiology (a first control group with axonal neuropathies and thus no ataxia in the foreground, a second group with ataxiating neuropathies : (anti-MAG neuropathy, neuronopathies of autoimmune origin) and a healthy control group without neuropathy).
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
jerky pursuits | Baseline, Day 0
  Comparison of video oculography results (saccadic pursuits) of patients with a diagnosis of CANVAS with those of the other groups
gaze evoked nystagmus | Baseline, Day 0
  Comparison of video oculography results (gaze evoked nystagmus) of patients with a diagnosis of CANVAS with those of the other groups
down beat nystagmus | Baseline, Day 0
  Comparison of video oculography results (down beat nystagmus) of patients with a diagnosis of CANVAS with those of the other groups
rebound nystagmus | Baseline, Day 0
  Comparison of video oculography results (rebound nystagmus) of patients with a diagnosis of CANVAS with those of the other groups

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, Choisir Une Région, France

REFERENCES:
- [Result] Fabri G, Brandi G, Altieri A, Bernardini P, Di Donna V, Falappa PG. [Analysis and the respiratory risks in a cement plant]. Ann Ist Super Sanita. 1981;17(3):581-6. No abstract available. Italian. PMID 6918204
- [Result] Weber KP, MacDougall HG, Halmagyi GM, Curthoys IS. Impulsive testing of semicircular-canal function using video-oculography. Ann N Y Acad Sci. 2009 May;1164:486-91. doi: 10.1111/j.1749-6632.2008.03730.x. PMID 19645955
- [Result] Larrazabal AJ, Garcia Cena CE, Martinez CE. Video-oculography eye tracking towards clinical applications: A review. Comput Biol Med. 2019 May;108:57-66. doi: 10.1016/j.compbiomed.2019.03.025. Epub 2019 Mar 30. PMID 31003180
- [Result] Gorges M, Pinkhardt EH, Kassubek J. Alterations of eye movement control in neurodegenerative movement disorders. J Ophthalmol. 2014;2014:658243. doi: 10.1155/2014/658243. Epub 2014 May 18. PMID 24955249
- [Result] Szmulewicz DJ, Waterston JA, MacDougall HG, Mossman S, Chancellor AM, McLean CA, Merchant S, Patrikios P, Halmagyi GM, Storey E. Cerebellar ataxia, neuropathy, vestibular areflexia syndrome (CANVAS): a review of the clinical features and video-oculographic diagnosis. Ann N Y Acad Sci. 2011 Sep;1233:139-47. doi: 10.1111/j.1749-6632.2011.06158.x. PMID 21950986
- [Result] Cortese A, Reilly MM, Houlden H. RFC1 CANVAS / Spectrum Disorder. 2020 Nov 25. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK564656/ PMID 33237689
- [Result] Szmulewicz DJ, Waterston JA, Halmagyi GM, Mossman S, Chancellor AM, McLean CA, Storey E. Sensory neuropathy as part of the cerebellar ataxia neuropathy vestibular areflexia syndrome. Neurology. 2011 May 31;76(22):1903-10. doi: 10.1212/WNL.0b013e31821d746e. PMID 21624989